CLINICAL TRIAL: NCT01757756
Title: A Phase 1 Placebo-Controlled Study To Assess The Safety, Tolerability, Pharmacokinetics And Effect On Midazolam Pharmacokinetics Of Multiple Oral Doses Of PF-05175157 In Otherwise Healthy Overweight And Obese Subjects
Brief Title: Multiple Dose Safety Toelrability, Pharmacokinetics and Midazolam Interaction In Healthy Overweight And Obese Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: Single | Purpose: Basic Science
Other Study IDs: B1731017
Record Dates: First submitted 2012-10-23; First posted 2012-12-31 (Estimated); Last update posted 2012-12-31 (Estimated); Status verified 2012-12

CONDITIONS: Diabetes Mellitus; Diabetes Mellitus, Type 2; Glucose Metabolism Disorders
MeSH Terms: conditions — Diabetes Mellitus; Diabetes Mellitus, Type 2; Glucose Metabolism Disorders | interventions — Midazolam

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (1):
- Arm Label Pf-05175157, placebo, midazolam (Experimental)
  Interventions: Drug: Pf-05175157; Drug: placebo; Drug: midazolam

INTERVENTIONS:
Drug: Pf-05175157 — 200-mg administered twice daily for 14 days
Drug: placebo — placebo administered twice daily for 14 days
Drug: midazolam — midazolam 3-mg admistered as single doses on Day 0 and Day 11.

SUMMARY:
This study is designed to assess the safety, tolerability and pharmacokinetics of multiple oral 200-mg doses of Pf-05175157 administered twice daily for 14 days in healthy overweight and obese subjects.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male and/or female subjects between the ages of 18 and 55 years, inclusive (Healthy is defined as no clinically relevant abnormalities identified by a detailed medical history, full physical examination, including blood pressure and pulse rate measurement, 12 lead ECG and clinical laboratory tests).
* Body Mass Index (BMI) of 25 to 35 kg/m2 inclusive; and a total body weight >50 kg (110 lbs).
* Subjects who are willing and able to comply with scheduled visits, treatment plan, laboratory tests, and other study procedures.

Exclusion Criteria:

* Evidence or history of clinically significant hematological, renal, endocrine, pulmonary, gastrointestinal, cardiovascular, hepatic, psychiatric, neurologic, or allergic disease (including drug allergies, but excluding untreated, asymptomatic, seasonal allergies at time of dosing).
* Evidence or history of any chronic ongoing or current pulmonary disease.
* History of smoking in the past 5 years and a history of smoking more than 10 pack years, or history or evidence of habitual use of other (non smoked) tobacco or nicotine containing products. Active ocular disease including infection, glaucoma, seasonal allergies, dry eye symptoms or retinal/optic nerve disease.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2012-10; Primary Completion 2012-11 (Actual); Study Completion 2012-11 (Actual)

PRIMARY OUTCOMES:
Maximum Observed Plasma Concentration (Cmax) | 0, 0.5, 1, 2, 3, 4, 6, 8, 10, 12 hrs postdose
Area Under the Curve from Time Zero to end of dosing interval (AUCtau) | 0, 0.5, 1, 2, 3, 4, 6, 8, 10, 12 hrs postdose
Time to Reach Maximum Observed Plasma Concentration (Tmax) | 0, 0.5, 1, 2, 3, 4, 6, 8, 10, 12 hrs postdose
Maximum Observed Plasma Concentration (Cmax) | 0, 0.5, 1, 2, 3, 4, 6, 8, 10, 12, 24, 36 and 48 hours postdose
Time to Reach Maximum Observed Plasma Concentration (Tmax) | 0, 0.5, 1, 2, 3, 4, 6, 8, 10, 12, 24, 36 and 48 hours postdose
Area Under the Curve from Time Zero to end of dosing interval (AUCtau) | 0, 0.5, 1, 2, 3, 4, 6, 8, 10, 12, 24, 36 and 48 hours postdose
Plasma Decay Half-Life (t1/2) | 0, 0.5, 1, 2, 3, 4, 6, 8, 10, 12, 24, 36 and 48 hours postdose
Apparent Volume of Distribution (Vz/F) | 0, 0.5, 1, 2, 3, 4, 6, 8, 10, 12, 24, 36 and 48 hours postdose
Apparent Oral Clearance (CL/F) | 0, 0.5, 1, 2, 3, 4, 6, 8, 10, 12, 24, 36 and 48 hours postdose
Accumulation Ratio (Rac) | 0, 0.5, 1, 2, 3, 4, 6, 8, 10, 12 hours postdose
Ae,tau | 0-12 hr
Ae% | 0-12 hr
Clr | 0-12 hr
Area Under the Curve From Time Zero to Last Quantifiable Concentration [AUC (0-t)] | 0, 0.5, 1, 2, 3, 4, 6, 8, 10, 12, 16, 24, 36 and 48 hours
Maximum Observed Plasma Concentration (Cmax) | 0, 0.5, 1, 2, 3, 4, 6, 8, 10, 12, 16, 24, 36 and 48 hours
Time to Reach Maximum Observed Plasma Concentration (Tmax) | 0, 0.5, 1, 2, 3, 4, 6, 8, 10, 12, 16, 24, 36 and 48 hours
Plasma Decay Half-Life (t1/2) | 0, 0.5, 1, 2, 3, 4, 6, 8, 10, 12, 16, 24, 36 and 48 hours
Area Under the Curve From Time Zero to Extrapolated Infinite Time [AUC (0 - 8)] | 0, 0.5, 1, 2, 3, 4, 6, 8, 10, 12, 16, 24, 36 and 48 hours
fasting triglycerides | 14 days
fasting LDL-cholesterol | 14 days
fasting total cholesterol | 14 days
fasting HDL cholesterol | 14 days

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Pfizer Investigational Site, South Miami, Florida, United States

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=B1731017&StudyName=Multiple%20Dose%20Safety%20Toelrability%2C%20Pharmacokinetics%20and%20Midazolam%20Interaction%20In%20Healthy%20Overweight%20And%20Obese%20Subjects